CLINICAL TRIAL: NCT00514904
Title: Non-inferiority of GSK Biologicals' Meningococcal Vaccine GSK134612 Versus Mencevax™ in Healthy Subjects Aged 2 Through 10 Years of Age
Brief Title: Non-Inferiority of Meningococcal Vaccine GSK134612 Versus Mencevax™ in 2-10 Year Old Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109495; 2012-000283-23 (EudraCT Number)
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-09

CONDITIONS: Infections, Meningococcal; Meningococcal Vaccines
Keywords: safety; meningococcal vaccine; immunogenicity
MeSH Terms: conditions — Meningococcal Infections

ARMS (2):
- Nimenrix Group (Experimental): Subjects received 1 dose of Nimenrix vaccine at Month 0. Nimenrix vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: Nimenrix
- Mencevax ACWY Group (Active Comparator): Subjects received 1 dose of Mencevax ACWY vaccine at Month 0. Mencevax ACWY vaccine was administered subcutaneously into the upper region of the non-dominant arm.
  Interventions: Biological: Mencevax

INTERVENTIONS:
Biological: Nimenrix — Single dose, intramuscular injection
  Other Names: Meningococcal vaccine GSK134612
  Arms: Nimenrix Group
Biological: Mencevax — Single dose, subcutaneous injection
  Arms: Mencevax ACWY Group

SUMMARY:
The purpose of this study is to demonstrate, in 2-10 year old subjects, the non-inferiority of meningococcal vaccine GSK134612 compared to licensed meningococcal vaccine Mencevax™.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Multicentre study with 2 treatment groups. Two blood samples will be taken, prior to and one month after vaccination, from the first 75% enrolled subjects per country independent of the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents or guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 2 and 10 years of age at the time of vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Previously completed routine childhood vaccinations to the best of his/her parents'/guardians' knowledge.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within one month of the dose of vaccine.
* Previous vaccination with meningococcal polysaccharide vaccine of serogroup A, C, W-135 and/or Y (for subjects below 6 years) or within the last five previous years (for subjects 6 years old or above).
* Previous vaccination with meningococcal polysaccharide conjugate vaccine of serogroups A, C, W-135 and/or Y.
* Previous vaccination with tetanus toxoid within the last month.
* History of meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary), including human immunodeficiency virus (HIV) infection, based on medical history and physical examination..
* History of reactions or allergic disease likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1504 (Actual)
Dates: Start 2007-09-18 (Actual); Primary Completion 2008-09-03 (Actual); Study Completion 2009-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- India (4):
  - GSK Investigational Site, Goa
  - GSK Investigational Site, Indore
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Vellore
- GSK Investigational Site, Beirut, Lebanon
- GSK Investigational Site, Sampaloc, Manila, Philippines
- GSK Investigational Site, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Memish ZA, Dbaibo G, Montellano M, Verghese VP, Jain H, Dubey AP, Bianco V, Van der Wielen M, Gatchalian S, Miller JM. Immunogenicity of a single dose of tetravalent meningococcal serogroups A, C, W-135, and Y conjugate vaccine administered to 2- to 10-year-olds is noninferior to a licensed-ACWY polysaccharide vaccine with an acceptable safety profile. Pediatr Infect Dis J. 2011 Apr;30(4):e56-62. doi: 10.1097/INF.0b013e31820e6e02. PMID 21278617
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 109495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109495 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1504 subjects were enrolled into the study, and 1501 of them were vaccinated.
Period: Overall Study
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Started | 1125 | 376
Completed | 1101 | 371
Not Completed | 24 | 5
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 21 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix Group | Mencevax ACWY Group | Total
Number analyzed (Participants) | 1125 | 376 | 1501
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.6 (2.49) | 5.5 (2.45) | 5.57 (2.48)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 526 | 175 | 701
  Male | 599 | 201 | 800
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central/ South Asian heritage, n(%) | 300 | 101 | 401
  Asian - Japanese heritage, n(%) | 2 | 1 | 3
  Asian - South East Asian heritage, n(%) | 597 | 199 | 796
  Native Hawaiian or other Pacific Islander, n(%) | 1 | 0 | 1
  White - Arabic/ North African heritage, n(%) | 221 | 74 | 295
  White - Caucasian/ European heritage, n(%) | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Vaccine Response to N. Meningitidis Serogroups A (MenA), MenC, MenY and MenW-135
Description: Vaccine response was defined as an rSBA titer of at least 1:32 in subjects initially seronegative (< 1:8) and as 4-fold increase in titer from pre- to post-vaccination in subjects initially seropositive (≥ 1:8).
Time Frame: One month after vaccination (Post-vaccination, study Month 1)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available and for whom assay results were available for antibodies against at least one study vaccine antigen component from the blood sample taken one month after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 723 | 240
Participants
  rSBA-MenA: number analyzed (Participants) | 594 | 192
  rSBA-MenA | 529 | 124
  rSBA-MenC: number analyzed (Participants) | 691 | 234
  rSBA-MenC | 664 | 210
  rSBA-MenW-135: number analyzed (Participants) | 691 | 236
  rSBA-MenW-135 | 673 | 195
  rSBA-MenY | 670 | 165
Statistical Analysis 1: Comparison: Nimenrix Group vs Mencevax ACWY Group; Test type: Non-Inferiority — Non-inferiority criterion: Lower limit [LL] of the 2-sided standardized asymptotic 95% confidence interval [CI] greater than or equal to (≥) -10%; Difference in percentage = 14.77, 95% CI 2-sided [10.26 to 20.23]
Statistical Analysis 2: Comparison: Nimenrix Group vs Mencevax ACWY Group; Test type: Non-Inferiority — Non-inferiority criterion: Lower limit [LL] of the 2-sided standardized asymptotic 95% confidence interval [CI] ≥-10%; Difference in percentage = 24.47, 95% CI 2-sided [17.52 to 31.87]
Statistical Analysis 3: Comparison: Nimenrix Group vs Mencevax ACWY Group; Test type: Non-Inferiority — Non-inferiority criterion: Lower limit [LL] of the 2-sided standardized asymptotic 95% confidence interval [CI] ≥-10%; Difference in percentage; Difference in percentage = 6.35, 95% CI 2-sided [2.68 to 11.08]
Statistical Analysis 4: Comparison: Nimenrix Group vs Mencevax ACWY Group; Test type: Non-Inferiority — Non-inferiority criterion: Lower limit [LL] of the 2-sided standardized asymptotic 95% confidence interval [CI] ≥-10%; Difference in percentage = 23.92, 95% CI 2-sided [18.02 to 30.3]

2. Primary Outcome: Number of Subjects With Grade 3 General Symptoms (Solicited and Unsolicited)
Description: Grade 3 symptom was defined as symptom that prevented normal, everyday activities.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 1125 | 376
Participants | 10 | 1
Statistical Analysis 1: Comparison: Nimenrix Group vs Mencevax ACWY Group; Test type: Non-Inferiority — Criterion for assessment: upper limit of the two-sided standardized asymptotic 95% confidence interval (CI) for the ratio between Nimenrix Group and Mencevax ACWY Group being lower than or equal to the pre-defined clinical limit ratio of 3.0 in the percentage of subjects with any grade 3 general symptoms; p = 0.2202, Chi-squared; Risk Ratio (RR) = 3.34, 95% CI 2-sided [0.56 to 20.25]

3. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY) Titers Greater Than or Equal (≥) to the Cut-off Values
Description: The cut-off values for the rSBA titers were ≥ 1:8 and ≥ 1:128 respectively.
Time Frame: Pre vaccination (Month 0) and post vaccination (Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 742 | 250
Participants
  rSBA-MenA ≥ 1:8, M0: number analyzed (Participants) | 599 | 194
  rSBA-MenA ≥ 1:8, M0 | 491 | 162
  rSBA-MenA≥ 1:8, M1: number analyzed (Participants) | 739 | 247
  rSBA-MenA≥ 1:8, M1 | 739 | 246
  rSBA-MenA ≥ 1:128, M0: number analyzed (Participants) | 599 | 194
  rSBA-MenA ≥ 1:128, M0 | 476 | 155
  rSBA-MenA≥ 1:128, M1: number analyzed (Participants) | 739 | 247
  rSBA-MenA≥ 1:128, M1 | 739 | 246
  rSBA-MenC≥ 1:8, M0: number analyzed (Participants) | 692 | 237
  rSBA-MenC≥ 1:8, M0 | 224 | 77
  rSBA-MenC≥ 1:8, M1: number analyzed (Participants) | 742 | 248
  rSBA-MenC≥ 1:8, M1 | 738 | 241
  rSBA-MenC ≥ 1:128 M0: number analyzed (Participants) | 692 | 237
  rSBA-MenC ≥ 1:128 M0 | 157 | 51
  rSBA-MenC ≥ 1:128 M1: number analyzed (Participants) | 742 | 248
  rSBA-MenC ≥ 1:128 M1 | 736 | 234
  rSBA-MenW-135 ≥ 1:8, M0: number analyzed (Participants) | 693 | 237
  rSBA-MenW-135 ≥ 1:8, M0 | 455 | 152
  rSBA-MenW-135 ≥ 1:8, M1 | 742 | 245
  rSBA-MenW-135. ≥ 1:128 M0: number analyzed (Participants) | 693 | 237
  rSBA-MenW-135. ≥ 1:128 M0 | 389 | 133
  rSBA-MenW-135 ≥ 1:128 M1 | 742 | 245
  rSBA-MenY ≥ 1:8, M0: number analyzed (Participants) | 725 | 241
  rSBA-MenY ≥ 1:8, M0 | 630 | 198
  rSBA-MenY ≥ 1:8, M1 | 742 | 248
  rSBA-MenY≥ 1:128 M0: number analyzed (Participants) | 725 | 241
  rSBA-MenY≥ 1:128 M0 | 590 | 188
  rSBA-MenY ≥ 1:128 M1 | 742 | 246

4. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers
Description: Antibody titers were expressed as geometric mean titers (GMTs).
Time Frame: Pre vaccination (Month 0) and post vaccination (Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 742 | 250
Titer
  rSBA-MenA, M0: number analyzed (Participants) | 599 | 194
  rSBA-MenA, M0 | 219.1 [186.5 to 257.4] | 227.7 [172.9 to 299.9]
  rSBA-MenA, M1: number analyzed (Participants) | 739 | 247
  rSBA-MenA, M1 | 6343.3 [5998.3 to 6708.1] | 2283.2 [2022.6 to 2577.3]
  rSBA-MenC, M0: number analyzed (Participants) | 692 | 237
  rSBA-MenC, M0 | 14.5 [12.5 to 16.7] | 14.2 [11.1 to 18.1]
  rSBA-MenC, M1: number analyzed (Participants) | 742 | 248
  rSBA-MenC, M1 | 4813.1 [4342.1 to 5335.3] | 1317 [1042.9 to 1663.3]
  rSBA-MenW-135, M0: number analyzed (Participants) | 693 | 237
  rSBA-MenW-135, M0 | 80.1 [67.4 to 95.3] | 68.8 [51.3 to 92.3]
  rSBA-MenW-135, M1 | 11543.2 [10872.7 to 12255.1] | 2157.8 [1815.2 to 2565.1]
  rSBA-MenY, M0: number analyzed (Participants) | 725 | 241
  rSBA-MenY, M0 | 310 [268.8 to 357.3] | 241.7 [185.3 to 315.3]
  rSBA-MenY, M1 | 10825.1 [10232.7 to 11451.7] | 2613.1 [2236.9 to 3052.5]

5. Secondary Outcome: Number of Subjects With Anti-tetanus Toxoid (Anti-TT) Concentrations Greater Than or Equal to (≥) the Cut-off Values
Description: The cut-off values for anti-TT concentrations were ≥ 0.1 international units per milliliter (IU/mL) and ≥ 1.0 IU/mL respectively.
Time Frame: Pre vaccination (Month 0) and post vaccination (Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 743 | 250
Participants
  Anti-TT ≥ 0.1 IU/mL, M0 | 635 | 220
  Anti-TT ≥ 0.1 IU/mL, M1: number analyzed (Participants) | 740 | 249
  Anti-TT ≥ 0.1 IU/mL, M1 | 733 | 218
  Anti-TT ≥ 1.0 IU/mL, M0 | 296 | 107
  Anti-TT ≥1.0 IU/mL, M1: number analyzed (Participants) | 740 | 249
  Anti-TT ≥1.0 IU/mL, M1 | 720 | 107

6. Secondary Outcome: Anti-tetanus Toxoid (Anti-TT) Antibody Concentrations
Description: Antibody concentrations were expressed as geometric mean concentrations (GMCs)
Time Frame: Pre vaccination (Month 0) and post vaccination (Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 743 | 250
Titer
  Anti-TT, M0 | 0.65 [0.577 to 0.731] | 0.744 [0.609 to 0.908]
  Anti-TT, M1: number analyzed (Participants) | 740 | 249
  Anti-TT, M1 | 21.731 [19.821 to 23.825] | 0.709 [0.581 to 0.866]

7. Secondary Outcome: Number of Subjects With Anti-polysaccharide (Anti-PS) Concentrations Greater Than or Equal to (≥) the Cut-off Values
Description: The cut-off values for anti-PS concentrations were ≥ 0.3 microgram per milliliter (μg/mL) and ≥ 2.0 μg/mL respectively for the anti- PSA, anti-PSC, anti-PSW-135 and anti-PSY antibodies respectively. One half of the subjects (50%, randomized) of the ATP cohort for immunogenicity was tested for anti-PSA and anti-PSC and the other half for anti-PSW-135 and anti-PSY.
Time Frame: Pre vaccination (Month 0) and post vaccination, (Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 370 | 128
Participants
  Anti-PSA ≥ 0.3 μg/mL, M0: number analyzed (Participants) | 354 | 124
  Anti-PSA ≥ 0.3 μg/mL, M0 | 154 | 41
  Anti-PSA ≥ 0.3 μg/mL, M1 | 369 | 126
  Anti-PSA ≥ 2.0 μg/mL, M0: number analyzed (Participants) | 354 | 124
  Anti-PSA ≥ 2.0 μg/mL, M0 | 59 | 12
  Anti-PSA ≥ 2.0 μg/mL, M1 | 368 | 123
  Anti-PSC ≥ 0.3 μg/mL, M0: number analyzed (Participants) | 368 | 127
  Anti-PSC ≥ 0.3 μg/mL, M0 | 29 | 7
  Anti-PSC ≥ 0.3 μg/mL, M1: number analyzed (Participants) | 366 | 127
  Anti-PSC ≥ 0.3 μg/mL, M1 | 365 | 127
  Anti-PSC ≥ 2.0 μg/mL, M0: number analyzed (Participants) | 368 | 127
  Anti-PSC ≥ 2.0 μg/mL, M0 | 12 | 2
  Anti-PSC ≥ 2.0 μg/mL M1: number analyzed (Participants) | 366 | 127
  Anti-PSC ≥ 2.0 μg/mL M1 | 363 | 125
  Anti-PSW-135 ≥ 0.3 μg/mL, M0: number analyzed (Participants) | 364 | 121
  Anti-PSW-135 ≥ 0.3 μg/mL, M0 | 18 | 11
  Anti-PSW-135 ≥ 0.3 μg/mL, M1: number analyzed (Participants) | 370 | 121
  Anti-PSW-135 ≥ 0.3 μg/mL, M1 | 368 | 121
  Anti-PSW-135 ≥ 2.0 μg/mL M0: number analyzed (Participants) | 364 | 121
  Anti-PSW-135 ≥ 2.0 μg/mL M0 | 5 | 2
  Anti-PSW-135 ≥ 2.0 μg/mL M1: number analyzed (Participants) | 370 | 121
  Anti-PSW-135 ≥ 2.0 μg/mL M1 | 353 | 112
  Anti-PSY ≥ 0.3 μg/mL, M0: number analyzed (Participants) | 368 | 121
  Anti-PSY ≥ 0.3 μg/mL, M0 | 28 | 16
  Anti-PSY ≥ 0.3 μg/mL, M1: number analyzed (Participants) | 370 | 122
  Anti-PSY ≥ 0.3 μg/mL, M1 | 369 | 122
  Anti-PSY ≥ 2.0 μg/mL, M0: number analyzed (Participants) | 368 | 121
  Anti-PSY ≥ 2.0 μg/mL, M0 | 11 | 4
  Anti-PSY ≥ 2.0 μg/mL, M1: number analyzed (Participants) | 370 | 122
  Anti-PSY ≥ 2.0 μg/mL, M1 | 362 | 118

8. Secondary Outcome: Anti-polysaccharide (Anti-PS) Antibody Concentrations
Description: Anti-PS concentrations were expressed as geometric mean concentrations (GMCs) and expressed in μg/mL. One half of the subjects (50%, randomized) of the ATP cohort for immunogenicity was tested for anti-PSA and anti-PSC and the other half for anti-PSW-135 and anti-PSY.
Time Frame: Pre vaccination (Month 0) and post vaccination (Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 370 | 128
μg/mL
  Anti-PSA, M0: number analyzed (Participants) | 354 | 124
  Anti-PSA, M0 | 0.4 [0.35 to 0.46] | 0.29 [0.24 to 0.36]
  Anti-PSA, M1 | 81.1 [71.34 to 92.2] | 25.43 [19.66 to 32.9]
  Anti-PSC, M0: number analyzed (Participants) | 368 | 127
  Anti-PSC, M0 | 0.18 [0.17 to 0.19] | 0.17 [0.15 to 0.18]
  Anti-PSC, M1: number analyzed (Participants) | 366 | 127
  Anti-PSC, M1 | 22.61 [20.24 to 25.25] | 25.69 [21.3 to 30.99]
  Anti-PSW-135, M0: number analyzed (Participants) | 364 | 121
  Anti-PSW-135, M0 | 0.17 [0.16 to 0.18] | 0.17 [0.16 to 0.19]
  Anti-PSW-135, M1: number analyzed (Participants) | 370 | 121
  Anti-PSW-135, M1 | 12.8 [11.32 to 14.48] | 13.85 [10.93 to 17.53]
  Anti-PSY, M0: number analyzed (Participants) | 368 | 121
  Anti-PSY, M0 | 0.18 [0.17 to 0.2] | 0.2 [0.17 to 0.23]
  Anti-PSY, M1: number analyzed (Participants) | 370 | 122
  Anti-PSY, M1 | 19.26 [17.1 to 21.69] | 22.71 [18.13 to 28.46]

9. Secondary Outcome: Number of Subjects Less Than (<) 6 Years of Age With Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as occurrence of any local symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects for whom data were available and with the symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 575 | 188
Participants
  Any Pain | 104 | 39
  Any Redness | 82 | 31
  Any Swelling | 31 | 15

10. Secondary Outcome: Number of Subjects ≥ 6 Years of Age With Solicited Local Symptoms
Description: as for outcome 9
Time Frame: During the 4-day (Days 0-3) follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and with the symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 542 | 186
Participants
  Any Pain | 105 | 50
  Any Redness | 107 | 36
  Any Swelling | 54 | 16

11. Secondary Outcome: Number of Subjects < 6 Years of Age With Solicited General Symptoms
Description: Solicited general symptoms assessed were drowsiness, fever (measured orally and temperature ≥ 37.5°C ), irritability and loss of appetite. Any was defined as incidence of any general symptom regardless of intensity grade or relationship to vaccination.
Time Frame: During the 4-day (Days 0-3) follow-up period after vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 575 | 188
Participants
  Any Drowsiness | 34 | 5
  Fever ≥ 37.5°C | 50 | 12
  Any Irritability | 31 | 6
  Any Loss of apptite | 35 | 6

12. Secondary Outcome: Number of Subjects ≥ 6 Years of Age With Solicited General Symptoms
Description: Solicited general symptoms assessed were fatigue, fever (measured orally and temperature ≥ 37.5°C ), gastrointestinal and headache. Any was defined as incidence of any general symptom regardless of intensity grade or relationship to vaccination.
Time Frame: During the 4-day (Days 0-3) follow-up period after vaccination
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 542 | 186
Participants
  Any Fatigue | 33 | 19
  Fever ≥ 37.5°C | 48 | 19
  Any Gastrointestinal | 25 | 15
  Any Headache | 51 | 19

13. Secondary Outcome: Number of Subjects Reporting Specific Adverse Events (AEs)
Description: Specific AEs include: rash; new onset of chronic illness(es) (NOCI) and/ or conditions prompting emergency room (ER) visits or non-routine physician office visits.
Time Frame: From Day 0 up to 6 months after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 1125 | 376
Participants
  Rash (es) | 45 | 16
  NOCI (s) | 3 | 1
  ER visit (s) | 15 | 4

14. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Symptoms
Description: Unsolicited symptom covers any symptom reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Up to one month (Day 0-Day 30) after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 1125 | 376
Participants | 198 | 75

15. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability /incapacity or are a congenital anomaly/ birth defect in the offspring of a study subject.
Time Frame: From Day 0 up to 6 months after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 1125 | 376
Participants | 15 | 7

ADVERSE EVENTS:
Time Frame: Serious adverse events: from Day 0 up to 6 months after vaccination. Solicited symptoms: during the 4-day (Day 0-Day 3) follow-up period after vaccination.
Description: The solicited local and general symptoms were only collected for those subjects who filled-in their symptom sheets.
Arm/Group | Nimenrix Group | Mencevax ACWY Group
All-Cause Mortality (participants affected / at risk) | 0/1125 | 0/376
Serious Adverse Events (participants affected / at risk) | 15/1125 | 7/376
Other Adverse Events (participants affected / at risk) | 416/1125 | 155/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix Group (N=1125) | Mencevax ACWY Group (N=376)
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Hyperchlorhydria (Skin and subcutaneous tissue disorders) | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Typhoid fever (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 3 | 1
Dengue fever (Infections and infestations) | 2 | 0
Otitis media (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 2 | 0
Amoebic dysentery (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Parasitic gastroenteritis (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nimenrix Group (N=1125) | Mencevax ACWY Group (N=376)
Pain (< 6 years of age) (General disorders) | 104/575 | 39/188 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects < 6 years of age.
Redness (< 6 years of age) (General disorders) | 82/575 | 31/188 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects < 6 years of age.
Swelling (< 6 years of age) (General disorders) | 31/575 | 15/188 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects 2-5 years of age.
Pain (≥ 6 years of age) (General disorders) | 105/575 | 50/188 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects ≥ 6 years of age.
Redness (≥ 6 years of age) (General disorders) | 107/542 | 36/186 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects ≥ 6 years of age.
Swelling (≥ 6 years of age) (General disorders) | 54/542 | 16/186 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects ≥ 6 years of age.
Drowsiness (General disorders) | 34/575 | 5/188 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects < 6 years of age.
Fever (Orally) (< 6 years of age) (General disorders) | 50/575 | 12/188 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects < 6 years of age.
Irritability (General disorders) | 31/575 | 6/188 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects < 6 years of age.
Loss of appetite (General disorders) | 35/575 | 6/188 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects < 6 years of age.
Fatigue (General disorders) | 33/542 | 19/186 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects ≥ 6 years of age.
Fever (Orally) (≥ 6 years of age) (General disorders) | 48/542 | 19/186 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects ≥ 6 years of age.
Gastrointestinal (General disorders) | 25/542 | 15/186 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects ≥ 6 years of age.
Headache (General disorders) | 51/542 | 19/186 — Assessed during the 4-day (Days 0-3) post-vaccination period in subjects ≥ 6 years of age.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.